CLINICAL TRIAL: NCT01481714
Title: Phase IV, Prospective, Randomized Study Comparing Preparation the Day Before and Split-dose Regimen With Sodium Picosulphate/Magnesium Citrate for Morning Colonoscopies
Brief Title: Efficacy and Safety of Split-dose Citrafleet Administered From 2 to 6 Hours Before Morning Colonoscopies
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Infante, Javier Molina, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CITRA-SPLIT
Record Dates: First submitted 2011-11-25; First posted 2011-11-29 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Bowel Cleansing; Colonoscopy
Keywords: Sodium picosulphate; Split-dose; Bowel cleansing; colonoscopy; Degree of bowel cleansing during colonoscopy
MeSH Terms: interventions — picosulfate sodium; Citric Acid; Magnesium Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium Picosulphate preparation the day before (Active Comparator): Preparation the day before of the procedure using sodium picosulphate:
  * A sachet mixed with 250 mL of water at 18:00 pm
  * A sachet mixed with 250 mL of water at 21:00 pm
  * A minimum of 4 litres of fluid were recommended throughout the preparation
  Interventions: Drug: Sodium picosulphate, magnesium oxid and citric acid
- Split-dose sodium picosulphate preparation (Experimental): The day before the procedure:
  - A sachet mixed with 250 mL of water at 18:00 pm, followed by 2 litres of clear liquids
  The day of the procedure:
  * A sachet administered at 5:45 am, followed by 1,5 litres of fluid intake up to 7 am for colonoscopies scheduled from 9 to 11 am.
  * A sachet administered at 6:45 am, followed by 1,5 litres of fluid intake up to 8 for colonoscopies scheduled after 11 am.
  Interventions: Drug: Sodium picosulphate/magnesium oxide and citric acid

INTERVENTIONS:
Drug: Sodium picosulphate, magnesium oxid and citric acid — * A sachet mixed with 250 mL of water at 18:00 pm
  * A sachet mixed with 250 mL of water at 21:00 pm
  * A minimum of 4 litres of fluid were recommended throughout the preparation
  Arms: Sodium Picosulphate preparation the day before
Drug: Sodium picosulphate/magnesium oxide and citric acid — The day before the procedure:
  - A sachet mixed with 250 mL of water at 18:00 pm, followed by 2 litres of clear liquids
  The day of the procedure:
  * A sachet administered at 5:45 am, followed by 1,5 litres of fluid intake up to 7 am for colonoscopies scheduled from 9 to 11 am.
  * A sachet administered at 6:45 am, followed by 1,5 litres of fluid intake up to 8 for colonoscopies scheduled after 11 am.
  Arms: Split-dose sodium picosulphate preparation

SUMMARY:
An excellent bowel cleansing is mandatory to increase the diagnostic accuracy of colonoscopy. Failure to adequately cleanse the bowel for colonoscopy can lead to missed lesions, prolonged procedure duration and repeated procedures at earlier intervals. Emerging solid evidence is pointing out the need of switching from preparation the day before to regimens in which half or even more of the preparation is administered the same day of the procedure, which have extensively demonstrated to provide a significantly better cleansing, being well tolerated. Preparation can be fully administered the same day for afternoon procedures, whereas split-dose regimens fit better with morning colonoscopies. However, the ideal regimen for early morning colonoscopies is still to be elucidated. The second part of the preparation for these patients is usually recommended to be taken during sleeping time (2-3 am) on the belief that intake of fluids should be completely halted at least four hours prior to the colonoscopy procedure Sodium picosulphate is a unique orange-flavoured cleansing agent dosed as two powder sachets. Mayor advantages in comparison with current alternatives are relatively small volumes (each sachet is mixed with only 150-250 mL of water) and a more pleasant taste. It provides similar bowel cleansing than sodium phosphate and polyethylene glycol solutions administered the day before. Nonetheless, focus on split-dose regimens has been set on several polyethylene glycol (either high-volume or low-volume) regimens, but no data are available for split-dose sodium-picosulphate regarding colonoscopy in adults.

The aim of the study is to evaluate the efficacy and safety of a sodium-picosulphate low-volume split-dose regimen, in which the second-half of the preparation and fluids intake are allowed until 2 hours for early morning colonoscopies and until 2-6 hours for morning colonoscopies, comparing this split-dose regimen with standard cleansing the day before with sodium picosulphate/magnesium citrate.

DETAILED DESCRIPTION:
Justification of the study:

Several split-dose bowel cleansing regimens have raised over the last decade aiming to substitute standard preparation the day before. These split-dose regimens (based on sodium phosphate and polyethylene glycol solutions) have demonstrated better cleansing scores, so it is probably more important the time that preparation is given rather than the type of solution. However, the time to administer the second half of the solution in split-dose regimens for morning colonoscopies remains controversial. A major concern of split-dose regimens is the risk of aspiration pneumonia during sedation if liquids have been administered quite close to the procedure. As such, the second part of the preparation is usually given early in the morning (2-3 am) in order to have a safety-period of at least four hours prior to the colonoscopy. However, this is quite disturbing for patients and may hamper the adherence to further colonoscopies. Furthermore, On the other hand, no study addressing the role of split-dose Citrafleet has been published to date

Therefore it is necessary to make a controlled clinical trial to directly compare "the day before" and " split-dose" regimens with Citrafleet for morning colonoscopies. In order to maximize the efficacy of the split-dose regimens, the time period between fluids intake and the colonoscopy will be shortened up up to 2 hours for morning colonoscopies scheduled from 9 to 11 am and up to 3 hours for that scheduled after 11 am. The results of this study will conclude whether there is still room for improvement in bowel cleansing for morning colonoscopies, using more palatable low-volume solutions without interrupting sleep time.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing routine elective colonoscopy

Exclusion Criteria:

* pregnant or lactating women
* age less than 18 years
* significant gastroparesis or gastric outlet obstruction or ileus
* known or suspected bowel obstruction or perforation
* phenylketonuria or glucose-6-phosphate dehydrogenase deficiency
* severe chronic renal failure (creatinine clearance < 30 mL/minute)
* severe congestive heart failure (New York Heart Association [NYHA] class III or IV)
* dehydration
* severe acute inflammatory disease
* compromised swallowing reflex or mental status
* uncontrolled hypertension (systolic blood pressure > 170 mm Hg ad/or diastolic blood pressure > 100 mm Hg)
* toxic colitis
* megacolon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-03 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Degree of bowel cleansing (Boston Scale 0-3) in each anatomical segment of the colon | 4 months
  Boston Scale: 3: excellent; 2: good ; 1: fair; 0: poor. Anatomical segments of the colon: rectum, sigmoid colon, descending colon, transverse colon, ascending colon and cecum

SECONDARY OUTCOMES:
Rate of aspiration bronchopneumonia | 4 months
Adenoma detection rate | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Javier Molina-Infante, MD, Principal Investigator — Hospital San Pedro de Alcantara, Caceres, Spain
Locations (1):
- Hospital San Pedro de Alcantara, Cáceres, Caceres, Spain

REFERENCES:
- [Background] Hoy SM, Scott LJ, Wagstaff AJ. Sodium picosulfate/magnesium citrate: a review of its use as a colorectal cleanser. Drugs. 2009;69(1):123-36. doi: 10.2165/00003495-200969010-00009. PMID 19192941
- [Background] Love J, Bernard EJ, Cockeram A, Cohen L, Fishman M, Gray J, Morgan D. A multicentre, observational study of sodium picosulfate and magnesium citrate as a precolonoscopy bowel preparation. Can J Gastroenterol. 2009 Oct;23(10):706-10. doi: 10.1155/2009/385619. PMID 19826647
- [Background] Turner D, Benchimol EI, Dunn H, Griffiths AM, Frost K, Scaini V, Avolio J, Ling SC. Pico-Salax versus polyethylene glycol for bowel cleanout before colonoscopy in children: a randomized controlled trial. Endoscopy. 2009 Dec;41(12):1038-45. doi: 10.1055/s-0029-1215333. Epub 2009 Dec 4. PMID 19967619
- [Background] Hookey LC, Vanner SJ. Pico-salax plus two-day bisacodyl is superior to pico-salax alone or oral sodium phosphate for colon cleansing before colonoscopy. Am J Gastroenterol. 2009 Mar;104(3):703-9. doi: 10.1038/ajg.2008.167. Epub 2009 Feb 17. PMID 19223885
- [Background] Worthington J, Thyssen M, Chapman G, Chapman R, Geraint M. A randomised controlled trial of a new 2 litre polyethylene glycol solution versus sodium picosulphate + magnesium citrate solution for bowel cleansing prior to colonoscopy. Curr Med Res Opin. 2008 Feb;24(2):481-8. doi: 10.1185/030079908x260844. PMID 18179734
- [Background] Renaut AJ, Raniga S, Frizelle FA, Perry RE, Guilford L. A randomized controlled trial comparing the efficacy and acceptability of phospo-soda buffered saline (Fleet) with sodium picosulphate/magnesium citrate (Picoprep) in the preparation of patients for colonoscopy. Colorectal Dis. 2008 Jun;10(5):503-5. doi: 10.1111/j.1463-1318.2007.01383.x. Epub 2007 Sep 13. PMID 17868404
- [Background] Park SS, Sinn DH, Kim YH, Lim YJ, Sun Y, Lee JH, Kim JY, Chang DK, Son HJ, Rhee PL, Rhee JC, Kim JJ. Efficacy and tolerability of split-dose magnesium citrate: low-volume (2 liters) polyethylene glycol vs. single- or split-dose polyethylene glycol bowel preparation for morning colonoscopy. Am J Gastroenterol. 2010 Jun;105(6):1319-26. doi: 10.1038/ajg.2010.79. Epub 2010 May 18. PMID 20485282
- [Background] Matro R, Shnitser A, Spodik M, Daskalakis C, Katz L, Murtha A, Kastenberg D. Efficacy of morning-only compared with split-dose polyethylene glycol electrolyte solution for afternoon colonoscopy: a randomized controlled single-blind study. Am J Gastroenterol. 2010 Sep;105(9):1954-61. doi: 10.1038/ajg.2010.160. Epub 2010 Apr 20. PMID 20407434
- [Background] Seo EH, Kim TO, Kim TG, Joo HR, Park MJ, Park J, Park SH, Yang SY, Moon YS. Efficacy and tolerability of split-dose PEG compared with split-dose aqueous sodium phosphate for outpatient colonoscopy: a randomized, controlled trial. Dig Dis Sci. 2011 Oct;56(10):2963-71. doi: 10.1007/s10620-011-1772-1. Epub 2011 Jun 9. PMID 21656179
- [Background] Kilgore TW, Abdinoor AA, Szary NM, Schowengerdt SW, Yust JB, Choudhary A, Matteson ML, Puli SR, Marshall JB, Bechtold ML. Bowel preparation with split-dose polyethylene glycol before colonoscopy: a meta-analysis of randomized controlled trials. Gastrointest Endosc. 2011 Jun;73(6):1240-5. doi: 10.1016/j.gie.2011.02.007. PMID 21628016
- [Background] Huffman M, Unger RZ, Thatikonda C, Amstutz S, Rex DK. Split-dose bowel preparation for colonoscopy and residual gastric fluid volume: an observational study. Gastrointest Endosc. 2010 Sep;72(3):516-22. doi: 10.1016/j.gie.2010.03.1125. Epub 2010 Jun 19. PMID 20646700
- [Background] Di Palma JA, Rodriguez R, McGowan J, Cleveland Mv. A randomized clinical study evaluating the safety and efficacy of a new, reduced-volume, oral sulfate colon-cleansing preparation for colonoscopy. Am J Gastroenterol. 2009 Sep;104(9):2275-84. doi: 10.1038/ajg.2009.389. Epub 2009 Jul 7. PMID 19584830
- [Background] Gupta T, Mandot A, Desai D, Abraham P, Joshi A, Shah S. Comparison of two schedules (previous evening versus same morning) of bowel preparation for colonoscopy. Endoscopy. 2007 Aug;39(8):706-9. doi: 10.1055/s-2007-966375. PMID 17661245
- [Background] Longcroft-Wheaton G, Bhandari P. Same-day bowel cleansing regimen is superior to a split-dose regimen over 2 days for afternoon colonoscopy: results from a large prospective series. J Clin Gastroenterol. 2012 Jan;46(1):57-61. doi: 10.1097/MCG.0b013e318233a986. PMID 22064553